CLINICAL TRIAL: NCT06326021
Title: Optimised CD33 (FL-33) CAR T Therapy for Refractory/Relapsed Acute Myeloid Leukaemia：a Multi-center, Open-label, Non-randomised, Single-arm Phase Ⅰ Clinical Trial
Brief Title: Optimised CD33 (FL-33) CAR T Therapy for Refractory/Relapsed Acute Myeloid Leukaemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: The General Hospital of Western Theater Command (Other); Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai (Other); Shanghai Liquan Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-004
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Refractory/Relapsed Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous FL-33 CAR T (Experimental): Peripheral blood mononuclear cells for the production of FL-33 CAR T cells are collected from patients.
  Interventions: Drug: autologous FL-33 CAR T therapy
- Prior-HSCT donor-derived FL-33 CAR T (Experimental): Peripheral blood mononuclear cells for the production of FL-33 CAR T cells are collected from prior-HSCT donors.
  Interventions: Drug: prior-HSCT donor-derived FL-33 CAR T therapy
- Newly matched donor-derived FL33 CAR T (Experimental): Peripheral blood mononuclear cells for the production of FL-33 CAR T cells are collected from newly matched donors.
  Interventions: Drug: Newly matched donor-derived FL-33 CAR T therapy

INTERVENTIONS:
Drug: autologous FL-33 CAR T therapy — Autologous FL-33 CAR T cells are infused intravenously.
  Arms: Autologous FL-33 CAR T
Drug: prior-HSCT donor-derived FL-33 CAR T therapy — Prior-HSCT donor-derived FL-33 CAR T cells are infused intravenously.
  Arms: Prior-HSCT donor-derived FL-33 CAR T
Drug: Newly matched donor-derived FL-33 CAR T therapy — Newly matched donor-derived FL-33 CAR T cells are infused intravenously
  Arms: Newly matched donor-derived FL33 CAR T

SUMMARY:
This study is a multi-center, open-label, non-randomised, single-arm phaseⅠclinical trial to explore the safety and efficacy of FL-33 CAR T therapy for refractory/relapsed acute myeloid leukaemia. The primary endpoints are incidence and type of dose limiting toxicity within 21 days of CAR T infusion; total number, incidence and severity of adverse events (AE) 30 days after CAR T infusion. The secondary endpoints are total number, incidence and severity of AEs 30 days to 2 years after CAR T infusion; objective response rate (ORR), complete response rate (CR) and complete response with incomplete haematological recovery (CRi) by dose group at 15, 30 and 90 Days after CAR T Infusion; duration of response (DOR), progression-free survival (PFS), overall survival (OS); pharmacokinetic characteristics. The trial will use BOIN12 design to explore the optimal biological dose (OBD) of FL-33 CAR T cells for refractory/relapsed acute myeloid leukaemia. FL-33 CAR T is set at two dose levels: 5*10^5 (±20%) CAR-T cells/kg for dose 1 (DL-1) and 1*10^6 (±20%) CAR-T cells/kg for dose 2 (DL-2), and after the optimal biological dose (OBD) is determined in the dose exploration phase, the dose expansion phase will expand the trial by 6-12 cases at the OBD, enrolling up to 21-27 cases. Enrolment of more than 21 cases can be reported for analysis and the trial will be stopped when enrolment reaches 27 cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met all the inclusion criteria were eligible for enrolment.

  1. Patients diagnosed with primary resistance acute myeloid leukemia, tumour surface antigen CD33 expression, chemotherapy relapse, extramedullary relapse, persistent residual positivity or relapse/refractory after allogeneic haematopoietic stem cell transplantation;
  2. Age 1-70 years old;
  3. No severe allergies;
  4. Physical condition: 0-2 ECOG score;
  5. Expected survival ≥ 60 days;
  6. Bone marrow or cerebrospinal fluid tumour cells are positive for CD33 by flow cytometry assay or tumour tissues positive for CD33 by immunohistochemistry (CD33 determination of positivity: flow cytometry: >80% of tumour cells expressing CD33 and MFI similar to normal myeloid cells is considered as full positivity; tumour cells greater than 80% of expression of CD33 but MFI lower than the CD33 expression of normal myeloid cells by 1 log is considered as low expression (dim). Tumour cells with between 20-80% positive CD33 expression are partially expressed; Pathological immunohistochemistry: tumour cells>30% positive are considered to be positively expressed;
  7. Self-aware patients aged 19-70 years are required to voluntarily sign an informed consent form in writing; paediatric patients aged 1-7 years can be recruited after their legal representative (guardian) had signed an informed consent form; self-aware paediatric patients aged 8-18 years voluntarily sign an informed consent form in writing, and their legal representative (guardian) are required to sign an informed consent form in writing as well;
  8. Suitable and available allogeneic haematopoietic stem cell transplant donors are required, and allogeneic haematopoietic stem cell transplantation can be performed after receiving FL-33 CAR T treatment.

Exclusion Criteria:

* Patients who fulfil any of the following criteria may not be enrolled.

  1. Patients with history of allogeneic HSCT but PBMNC is not available from prior- transplant donor for preparation of CAR T cells and peripheral blood tumour load >30%; patients without history of allogeneic HSCT and peripheral blood tumour load >30%;
  2. Intracranial hypertension or cerebral impaired consciousness;
  3. Symptomatic heart failure or severe arrhythmia;
  4. Symptoms of severe respiratory failure;
  5. With other types of malignancy;
  6. Diffuse intravascular coagulation;
  7. Serum creatinine and/or urea nitrogen ≥ 1.5 times the normal value;
  8. With sepsis or other uncontrollable infection;
  9. Suffering from uncontrollable diabetes mellitus;
  10. Severe mental disorders;
  11. Have significant intracranial lesions on cranial MRI;
  12. Organ transplantation (excluding haematopoietic stem cell transplantation) history;
  13. Female patients (patients of childbearing potential) with positive blood HCG test;
  14. Hepatitis (including hepatitis B and C) and positive screening for AIDS and syphilis.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 21 days
  Incidence and type of dose-limiting toxicity(DLT) within 21 days of FL-33 CAR T infusion.
Adverse events (AEs) | 30 days
  Total number, incidence and severity of adverse events (AEs) within 30 days of FL-33 CAR T infusion.

SECONDARY OUTCOMES:
Long-term Adverse events (AEs) | From 30 days after FL-33 CAR T infusion to 2 years
  Total number, incidence and severity of AEs from 30 days to 2 years after FL-33 CAR T infusion will be recorded.
Objective Response Rate (ORR) | 15, 30, 90 days
  The assessment of ORR by dose group at 15, 30 and 90 Days after FL-33 CAR T infusion according to National Comprehensive Cancer Network (NCCN) Guidelines Version 1.2024 of Acute myeloid Leukemia.
Duration of response (DOR) | Up to 2 years
  DOR is defined as the date when CR or CRi response criteria are first met to the date of relapse or death caused by AML in the absence of documented relapse.
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the earliest date of occurrence from the first infusion of FL-33 CAR T cells back into the patient who achieved ORR to the earliest date of death from any cause after relapse or remission.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from FL-33 CAR T infusion to death due to any cause.
The persistence of FL-33 CAR T cells | Up to 2 years
  The persistence of FL-33 CAR T cells in cerebral spinal fluid (CSF) and peripheral blood (PB) will be measured by flowcytometry and quantitative polymerase chain reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Liquan Hospital, Shanghai, Shanghai Municipality
  - The General Hospital of Western Theater Command PLA, Chengdu, Sichuan
  - BeijingGoBroadH, Beijing